CLINICAL TRIAL: NCT03461016
Title: Randomized Clinical Trial of Smartphone-Based Exposure of Dental Anxiety
Brief Title: Smartphone-Based Exposure Treatment for Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Daniel W. McNeil, PhD, Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1506718933
Record Dates: First submitted 2018-02-16; First posted 2018-03-09 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Phobic Disorders; Dental Anxiety; Treatment Outcome
Keywords: Smartphones; Exposure Therapy; Dental Anxiety
MeSH Terms: conditions — Phobic Disorders | interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone-Based Exposure Therapy (Experimental): Participants assigned to the Smartphone-Based Exposure Therapy group will receive two weeks of exposure therapy via their smartphone. Participants will have the opportunity to receive up to 50 minutes of exposure video intervention daily for the two weeks.
  Interventions: Behavioral: Exposure Therapy
- Waitlist Control (No Intervention): Participants who have been randomly assigned to participate in the Waitlist Control group will not receive treatment; however, after the two weeks of no intervention, participants in this condition will be offered the same treatment as the treatment condition.

INTERVENTIONS:
Behavioral: Exposure Therapy — "Exposure therapy is a form of behavior therapy that is widely used to treat anxiety disorders, including specific phobia. It involves systematic and repeated confrontation with a feared stimulus. It works by (a) implosive therapy, habituation, in which repeated exposure reduces anxiety over time by a process of extinction; (b) disconfirming fearful predictions; and (c) increasing feelings of self-efficacy and mastery. In vivo exposure [is] a type of exposure therapy, generally used for treating individuals with phobias, obsessive compulsive disorder, and other anxiety disorders, in which the client directly experiences anxiety-provoking situations or stimuli in real-world conditions." (VandenBos, 2015)
  Arms: Smartphone-Based Exposure Therapy

SUMMARY:
Exposure therapy, including its self-directed forms, is effective for treatment of specific phobias. Nevertheless, there are issues with patient adherence in the use of exposure therapy, including its self-directed formats. Technological advancements, as with smartphones, may improve adherence to self-directed exposure therapy, perhaps due to exposure stimuli being more readily accessible. Thus, there is a need to examine how presenting phobic material on a smartphone might promote increased adherence in conducting self-directed exposure. Additionally, exposure can incorporate phobic material from different perspectives (i.e., first-person or third-person), which is one factor that may impact treatment effectiveness. Participants will be randomly assigned to a treatment or control condition, and complete a pre-assessment and then a post-assessment two weeks later. The assessment consists of a multimodal approach (e.g., self-report, physiological response, and overt behavior). Participants in the treatment condition will be instructed to watch a standard exposure video of a dental examination and prophylaxis three times daily for two weeks. One week of videos was shown in a first-person perspective and the same video will be shown in a third-person perspective for one week. The study can demonstrate the potential utility of smartphone-based self-directed exposure therapy for specific phobia.

DETAILED DESCRIPTION:
1. Recruitment efforts will be made in the community via advertisements and online advertisements (e.g., Craigslist, Facebook).
2. Prospective participants will contact the investigators via email or by calling the study phone number listed on the advertisements.
3. Once a participant indicates interest by contacting study personnel, a 5-minute screening interview will be conducted with the prospective participant using the screening questionnaire to ensure eligibility criteria are met. For those who do not qualify or agree to participate, the age and reason for non-qualification or declination to participate will be recorded; any other data will be destroyed by shredding or electronic shredding. For those who do qualify, name and contact information will be kept confidential and maintained in a locked room.
4. After written agreement to enlist in the study, participants are randomly assigned to group (i.e., treatment or control) by previously prepared sealed opaque envelopes.
5. Participants will complete the demographic questionnaire, the Dental Fear Survey, and the investigator will complete the specific phobia section of the ADIS-5 with the participant.
6. Then a Behavioral Avoidance Task will be conducted with the participants

   1. One-minute baseline, in which the participant sat quietly.
   2. Then nine dental-related steps will be completed each lasted 30 seconds, and a SUDS rating was collected at each step.
7. After completing the Behavioral Avoidance Task, the investigator provides a 15-minute demonstration to the participants.

   1. The control group watched a video on their smartphone about smartphone capabilities as an attention control.
   2. The treatment group was shown how to conduct self-directed exposure therapy and rate SUDS on their smartphone.

   i. The video is a typical preventive visit to the dentist, including walking into the dental office, being called back for treatment by the dental assistant, sitting in the dental chair, and seeing the hygienist perform a teeth cleaning.

   ii. The video is presented in a first and third person perspective, and the order is randomly assigned (e.g., view the first person perspective video during week 1 of treatment and then third person perspective during week 2 of treatment).
8. Researcher will model how to rate SUDS prior to watching the exposure video, how to access the exposure video, how to rate actual SUDS experienced during the video, and how to either continue to the next video or stop the exposure session.

   1. Participants are advised that watching the exposure video three times per day is the ideal, which may match the amount of exposure in a typical 50-minute treatment session.
   2. One time per day was the suggested minimum, and five times per day was the suggested maximum.
9. An email will be sent to participants in the treatment group daily to remind them to conduct the exposure session over the two weeks of treatment.

   1. Participants follow the link each day with their smartphones. Before each exposure video, participants rate expected distress on the SUDS. Then asked to watch a video depicting dental care-related material. After viewing the exposure video, participants rated actual distress experienced on the SUDS.
   2. The participants then are immediately prompted to watch the video again. If the participant chooses to watch the video again, the participant will do the same procedure of pre-rating anxiety, watching the video, and post-rating anxiety.
   3. Finally, participants are prompted to complete the procedure a third time. After completing the procedure three times, the participants are no longer prompted, however, they had the ability to complete the procedure up to two more times if they so desired.
10. One week after the pre-assessment, participants are contacted via telephone by the investigator to complete measures and schedule the post-assessment session.

    1. Participants in the control condition will complete the Dental Fear Survey
    2. Participants in the treatment condition will complete the Dental Fear Survey and the IGroup Presence Questionnaire.
11. Participants return for the post-assessment session at least two-weeks after the pre-assessment to complete questionnaires and conduct the Behavioral Avoidance Task again.

    1. Participants in the control condition will complete the Dental Fear Survey
    2. Participants in the treatment condition will complete the Dental Fear Survey, IGroup Presence Questionnaire, and Acceptance and Acceptability Rating Profile.

ELIGIBILITY:
Inclusion Criteria:

* fluency in the English language
* being 18 years of age or older
* own or have access to a smartphone
* have an e-mail account

Exclusion Criteria:

* Reporting a low level of discomfort with dental-related care (i.e., less than a rating of "somewhat" on a single-item dental fear question)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Dental Fear Survey (scale 20-item) | Change from Baseline to 14 days
  Participant self-report of dental care-related fear and anxiety, range of 20-100

SECONDARY OUTCOMES:
Change in Subjective Units of Distress (scale 1-item) | Change from Baseline to 14 days
  Participant self-report of Anxiety, scale of 0-100
Acceptability (scale 8-item) | 14 days
  Participant self-report of the acceptability of treatment, range of 1-48

OTHER OUTCOMES:
Change in Behavioral Avoidance Task behavior | Change from Baseline to 14 days
  Nine steps of a simulated a dental examination

CONTACTS AND LOCATIONS:
Overall Officials: Daneil W McNeil, PhD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] VandenBos, G. R. (Ed.) (2015). APA dictionary of psychology. Washington, DC: American Psychological Association.

DOCUMENTS (2):
  • Study Protocol (2016-03-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT03461016/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT03461016/SAP_001.pdf